CLINICAL TRIAL: NCT05495685
Title: Pancreatic Cancer Detection by Liquid Biopsy in Peripheral Blood: A Prospective Study
Brief Title: iDentification and vAlidation Model of Liquid biopsY Based cfDNA Methylation and pRotEin biomArKers for Pancreatic Cancer (DAYBREAK Study)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Changhai Hospital (Other)
Collaborators: Guangzhou Burning Rock Bioengineering Ltd. (Industry)
Responsible Party: Principal Investigator, Guo ShiWei, Associated Professor at the Institute of Pancreatic Surgery, Changhai Hospital
Other Study IDs: CHEC2022-030
Record Dates: First submitted 2022-08-09; First posted 2022-08-10 (Actual); Last update posted 2022-08-10 (Actual); Status verified 2022-08

CONDITIONS: Cancer
Keywords: pancreatic cancer; liquid biopsy; cell-free DNA (cfDNA) methylation; whole blood miRNA; others
MeSH Terms: conditions — Neoplasms; Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cancer arm: Participants with new diagnosis of pancreatic cancer, from whom a blood sample will be collected.
- Benign disease arm: Participants with benign pancreatic diseases, from whom a blood sample will be collected.

SUMMARY:
DAYBREAK is a prospective, multi-omics, observational study aimed at early detecting pancreatic cancer by combined assays for biomarkers of cfDNA methylation, serum protein markers, blood miRNA markers and others, in which of 450 participants will be enrolled. The development and validation of the model will be conducted in participants with early stage cancers and benign disease through a two-stage approach. The sensitivity and specificity of the model in pancreatic cancer early detection will be evaluated.

ELIGIBILITY:
Inclusion Criteria for Cancer Arm Participants:

* Able to provide a written informed consent.
* Able to provide sufficient and qualified blood samples for study tests.
* No prior or undergoing cancer treatment (local or systematic) with either of the following:
* A. Pathologically confirmed cancer diagnosis within 42 days prior to the study blood draw.
* B. High suspicious for cancer diagnosis by radiological or other routine clinical assessments, with confirmed cancer diagnosis through biopsy or surgical resection within 42 days after study blood draw.

Exclusion Criteria for Cancer Arm Participants:

* Insufficient qualified blood sample for study test.
* During pregnancy or lactation.
* Recipient of organ transplant or prior non-autologous (allogeneic) bone marrow or stem cell transplant.
* Recipient of blood transfusion within 30 days prior to study blood draw.
* With other known malignant tumors or multiple primary tumors.

Inclusion Criteria for Benign Disease Arm Participants:

* Able to provide a written informed consent.
* Able to provide sufficient and qualified blood samples for study tests.
* Have either of the following:
* A. Pathological confirmed diagnosis of benign diseases within 90 days prior to the study blood draw, with no prior treatment such as surgical resection.
* B. High suspicious for benign diseases diagnosis by radiological or other routine clinical assessments, with confirmed benign diseases diagnosis within 42 days after study blood draw.

Exclusion Criteria for Benign Disease Arm Participants:

* Insufficient qualified blood sample for study test.
* During pregnancy or lactation.
* Recipient of organ transplant or prior non-autologous (allogeneic) bone marrow or stem cell transplant.
* Recipient of blood transfusion within 30 days prior to study blood draw.
* Recipients of any anti-cancer therapy within 30 days prior to study blood draw, due to diseases other than cancer

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Eligible participants will be recruited from medical centers and assigned into two arms, including participants with new diagnosis of malignancy or corresponding benign disease.
Sampling Method: Non-Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2022-03-24 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
The sensitivity and specificity of multi-cancer early detection by the combined model in cancer arm and benign disease arm | 12 months

SECONDARY OUTCOMES:
The difference of sensitivity and specificity in pancreatic cancer participants at different clinical stages. | 12 months
Sensitivity and specificity for detecting pancreatic cancer of a cfDNA methylation-based model, in combination with other biomarkers. | 12 months
Sensitivity and specificity for detecting pancreatic cancer of a the protein panel-based model, in combination with other biomarkers. | 12 months
Sensitivity and specificity of the blood miRNA-based model in detecting pancreatic cancer. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Gang Jin, M.D., Study Chair — Department of general surgery, Changhai Hospital
Locations (1):
- Shanghai Changhai Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Steel N, Ford JA, Newton JN, Davis ACJ, Vos T, Naghavi M, Glenn S, Hughes A, Dalton AM, Stockton D, Humphreys C, Dallat M, Schmidt J, Flowers J, Fox S, Abubakar I, Aldridge RW, Baker A, Brayne C, Brugha T, Capewell S, Car J, Cooper C, Ezzati M, Fitzpatrick J, Greaves F, Hay R, Hay S, Kee F, Larson HJ, Lyons RA, Majeed A, McKee M, Rawaf S, Rutter H, Saxena S, Sheikh A, Smeeth L, Viner RM, Vollset SE, Williams HC, Wolfe C, Woolf A, Murray CJL. Changes in health in the countries of the UK and 150 English Local Authority areas 1990-2016: a systematic analysis for the Global Burden of Disease Study 2016. Lancet. 2018 Nov 3;392(10158):1647-1661. doi: 10.1016/S0140-6736(18)32207-4. Epub 2018 Oct 24. PMID 30497795
- [Background] Chen W, Zheng R, Baade PD, Zhang S, Zeng H, Bray F, Jemal A, Yu XQ, He J. Cancer statistics in China, 2015. CA Cancer J Clin. 2016 Mar-Apr;66(2):115-32. doi: 10.3322/caac.21338. Epub 2016 Jan 25. PMID 26808342
- [Background] Smith RA, Andrews KS, Brooks D, Fedewa SA, Manassaram-Baptiste D, Saslow D, Brawley OW, Wender RC. Cancer screening in the United States, 2018: A review of current American Cancer Society guidelines and current issues in cancer screening. CA Cancer J Clin. 2018 Jul;68(4):297-316. doi: 10.3322/caac.21446. Epub 2018 May 30. PMID 29846940
- [Background] O'Neill RS, Stoita A. Biomarkers in the diagnosis of pancreatic cancer: Are we closer to finding the golden ticket? World J Gastroenterol. 2021 Jul 14;27(26):4045-4087. doi: 10.3748/wjg.v27.i26.4045. PMID 34326612
- [Background] Orntoft TF, Vestergaard EM, Holmes E, Jakobsen JS, Grunnet N, Mortensen M, Johnson P, Bross P, Gregersen N, Skorstengaard K, Jensen UB, Bolund L, Wolf H. Influence of Lewis alpha1-3/4-L-fucosyltransferase (FUT3) gene mutations on enzyme activity, erythrocyte phenotyping, and circulating tumor marker sialyl-Lewis a levels. J Biol Chem. 1996 Dec 13;271(50):32260-8. doi: 10.1074/jbc.271.50.32260. PMID 8943285
- [Background] Luo G, Jin K, Deng S, Cheng H, Fan Z, Gong Y, Qian Y, Huang Q, Ni Q, Liu C, Yu X. Roles of CA19-9 in pancreatic cancer: Biomarker, predictor and promoter. Biochim Biophys Acta Rev Cancer. 2021 Apr;1875(2):188409. doi: 10.1016/j.bbcan.2020.188409. Epub 2020 Aug 19. PMID 32827580
- [Background] Luo G, Guo M, Jin K, Liu Z, Liu C, Cheng H, Lu Y, Long J, Liu L, Xu J, Ni Q, Yu X. Optimize CA19-9 in detecting pancreatic cancer by Lewis and Secretor genotyping. Pancreatology. 2016 Nov-Dec;16(6):1057-1062. doi: 10.1016/j.pan.2016.09.013. Epub 2016 Sep 23. PMID 27692554
- [Background] Zhu G, Pei L, Xia H, Tang Q, Bi F. Role of oncogenic KRAS in the prognosis, diagnosis and treatment of colorectal cancer. Mol Cancer. 2021 Nov 6;20(1):143. doi: 10.1186/s12943-021-01441-4. PMID 34742312
- [Background] Bournet B, Selves J, Grand D, Danjoux M, Hanoun N, Cordelier P, Buscail L. Endoscopic ultrasound-guided fine-needle aspiration biopsy coupled with a KRAS mutation assay using allelic discrimination improves the diagnosis of pancreatic cancer. J Clin Gastroenterol. 2015 Jan;49(1):50-6. doi: 10.1097/MCG.0000000000000053. PMID 24798941
- [Background] Riva G, Pea A, Pilati C, Fiadone G, Lawlor RT, Scarpa A, Luchini C. Histo-molecular oncogenesis of pancreatic cancer: From precancerous lesions to invasive ductal adenocarcinoma. World J Gastrointest Oncol. 2018 Oct 15;10(10):317-327. doi: 10.4251/wjgo.v10.i10.317. PMID 30364837
- [Background] Kirkegard J, Mortensen FV, Cronin-Fenton D. Chronic Pancreatitis and Pancreatic Cancer Risk: A Systematic Review and Meta-analysis. Am J Gastroenterol. 2017 Sep;112(9):1366-1372. doi: 10.1038/ajg.2017.218. Epub 2017 Aug 1. PMID 28762376
- [Background] Basturk O, Hong SM, Wood LD, Adsay NV, Albores-Saavedra J, Biankin AV, Brosens LA, Fukushima N, Goggins M, Hruban RH, Kato Y, Klimstra DS, Kloppel G, Krasinskas A, Longnecker DS, Matthaei H, Offerhaus GJ, Shimizu M, Takaori K, Terris B, Yachida S, Esposito I, Furukawa T; Baltimore Consensus Meeting. A Revised Classification System and Recommendations From the Baltimore Consensus Meeting for Neoplastic Precursor Lesions in the Pancreas. Am J Surg Pathol. 2015 Dec;39(12):1730-41. doi: 10.1097/PAS.0000000000000533. PMID 26559377
- [Background] Hruban RH, Adsay NV, Albores-Saavedra J, Compton C, Garrett ES, Goodman SN, Kern SE, Klimstra DS, Kloppel G, Longnecker DS, Luttges J, Offerhaus GJ. Pancreatic intraepithelial neoplasia: a new nomenclature and classification system for pancreatic duct lesions. Am J Surg Pathol. 2001 May;25(5):579-86. doi: 10.1097/00000478-200105000-00003. PMID 11342768
- [Background] Luchini C, Capelli P, Scarpa A. Pancreatic Ductal Adenocarcinoma and Its Variants. Surg Pathol Clin. 2016 Dec;9(4):547-560. doi: 10.1016/j.path.2016.05.003. Epub 2016 Oct 12. PMID 27926359
- [Background] Sato N, Fukushima N, Hruban RH, Goggins M. CpG island methylation profile of pancreatic intraepithelial neoplasia. Mod Pathol. 2008 Mar;21(3):238-44. doi: 10.1038/modpathol.3800991. Epub 2007 Dec 21. PMID 18157091
- [Background] Gaujoux S, Chanson P, Bertherat J, Sauvanet A, Ruszniewski P. Hepato-pancreato-biliary lesions are present in both Carney complex and McCune Albright syndrome: comments on P. Salpea and C. Stratakis. Mol Cell Endocrinol. 2014 Jan 25;382(1):344-345. doi: 10.1016/j.mce.2013.10.020. Epub 2013 Oct 24. PMID 24161590
- [Background] Shi C, Klein AP, Goggins M, Maitra A, Canto M, Ali S, Schulick R, Palmisano E, Hruban RH. Increased Prevalence of Precursor Lesions in Familial Pancreatic Cancer Patients. Clin Cancer Res. 2009 Dec 15;15(24):7737-7743. doi: 10.1158/1078-0432.CCR-09-0004. PMID 19996207
- [Background] Ingkakul T, Sadakari Y, Ienaga J, Satoh N, Takahata S, Tanaka M. Predictors of the presence of concomitant invasive ductal carcinoma in intraductal papillary mucinous neoplasm of the pancreas. Ann Surg. 2010 Jan;251(1):70-5. doi: 10.1097/SLA.0b013e3181c5ddc3. PMID 20009749
- [Background] Fukushige S, Horii A. Road to early detection of pancreatic cancer: Attempts to utilize epigenetic biomarkers. Cancer Lett. 2014 Jan 28;342(2):231-7. doi: 10.1016/j.canlet.2012.03.022. Epub 2012 Mar 23. PMID 22450751
- [Background] Curradi M, Izzo A, Badaracco G, Landsberger N. Molecular mechanisms of gene silencing mediated by DNA methylation. Mol Cell Biol. 2002 May;22(9):3157-73. doi: 10.1128/MCB.22.9.3157-3173.2002. PMID 11940673
- [Background] Kim SG, Wu TT, Lee JH, Yun YK, Issa JP, Hamilton SR, Rashid A. Comparison of epigenetic and genetic alterations in mucinous cystic neoplasm and serous microcystic adenoma of pancreas. Mod Pathol. 2003 Nov;16(11):1086-94. doi: 10.1097/01.MP.0000094088.37888.A6. PMID 14614047
- [Background] Keane MG, Afghani E. A Review of the Diagnosis and Management of Premalignant Pancreatic Cystic Lesions. J Clin Med. 2021 Mar 19;10(6):1284. doi: 10.3390/jcm10061284. PMID 33808853
- [Background] Delpu Y, Hanoun N, Lulka H, Sicard F, Selves J, Buscail L, Torrisani J, Cordelier P. Genetic and epigenetic alterations in pancreatic carcinogenesis. Curr Genomics. 2011 Mar;12(1):15-24. doi: 10.2174/138920211794520132. PMID 21886451
- [Background] 岳铭, 徐海燕, 张晓飞, 王理伟. 胰腺炎--癌转化的表观遗传学研究进展. 肿瘤防治研究. 2021;48(3):219-223
- [Background] Natale F, Vivo M, Falco G, Angrisano T. Deciphering DNA methylation signatures of pancreatic cancer and pancreatitis. Clin Epigenetics. 2019 Sep 6;11(1):132. doi: 10.1186/s13148-019-0728-8. PMID 31492175
- [Background] Matsubayashi H, Canto M, Sato N, Klein A, Abe T, Yamashita K, Yeo CJ, Kalloo A, Hruban R, Goggins M. DNA methylation alterations in the pancreatic juice of patients with suspected pancreatic disease. Cancer Res. 2006 Jan 15;66(2):1208-17. doi: 10.1158/0008-5472.CAN-05-2664. PMID 16424060
- [Background] Chen M, Zhao H. Next-generation sequencing in liquid biopsy: cancer screening and early detection. Hum Genomics. 2019 Aug 1;13(1):34. doi: 10.1186/s40246-019-0220-8. PMID 31370908
- [Background] Moore LD, Le T, Fan G. DNA methylation and its basic function. Neuropsychopharmacology. 2013 Jan;38(1):23-38. doi: 10.1038/npp.2012.112. Epub 2012 Jul 11. PMID 22781841
- [Background] Guibert S, Weber M. Functions of DNA methylation and hydroxymethylation in mammalian development. Curr Top Dev Biol. 2013;104:47-83. doi: 10.1016/B978-0-12-416027-9.00002-4. PMID 23587238
- [Background] Widschwendter M, Jones A, Evans I, Reisel D, Dillner J, Sundstrom K, Steyerberg EW, Vergouwe Y, Wegwarth O, Rebitschek FG, Siebert U, Sroczynski G, de Beaufort ID, Bolt I, Cibula D, Zikan M, Bjorge L, Colombo N, Harbeck N, Dudbridge F, Tasse AM, Knoppers BM, Joly Y, Teschendorff AE, Pashayan N; FORECEE (4C) Consortium. Epigenome-based cancer risk prediction: rationale, opportunities and challenges. Nat Rev Clin Oncol. 2018 May;15(5):292-309. doi: 10.1038/nrclinonc.2018.30. Epub 2018 Feb 27. PMID 29485132
- [Background] Vogelstein B, Papadopoulos N, Velculescu VE, Zhou S, Diaz LA Jr, Kinzler KW. Cancer genome landscapes. Science. 2013 Mar 29;339(6127):1546-58. doi: 10.1126/science.1235122. PMID 23539594
- [Background] Guo S, Diep D, Plongthongkum N, Fung HL, Zhang K, Zhang K. Identification of methylation haplotype blocks aids in deconvolution of heterogeneous tissue samples and tumor tissue-of-origin mapping from plasma DNA. Nat Genet. 2017 Apr;49(4):635-642. doi: 10.1038/ng.3805. Epub 2017 Mar 6. PMID 28263317
- [Background] Johnson DA, Barclay RL, Mergener K, Weiss G, Konig T, Beck J, Potter NT. Plasma Septin9 versus fecal immunochemical testing for colorectal cancer screening: a prospective multicenter study. PLoS One. 2014 Jun 5;9(6):e98238. doi: 10.1371/journal.pone.0098238. eCollection 2014. PMID 24901436
- [Background] Church TR, Wandell M, Lofton-Day C, Mongin SJ, Burger M, Payne SR, Castanos-Velez E, Blumenstein BA, Rosch T, Osborn N, Snover D, Day RW, Ransohoff DF; PRESEPT Clinical Study Steering Committee, Investigators and Study Team. Prospective evaluation of methylated SEPT9 in plasma for detection of asymptomatic colorectal cancer. Gut. 2014 Feb;63(2):317-25. doi: 10.1136/gutjnl-2012-304149. Epub 2013 Feb 13. PMID 23408352
- [Background] Ilse P, Biesterfeld S, Pomjanski N, Wrobel C, Schramm M. Analysis of SHOX2 methylation as an aid to cytology in lung cancer diagnosis. Cancer Genomics Proteomics. 2014 Sep-Oct;11(5):251-8. PMID 25331797
- [Background] 肺癌筛查与管理中国专家共识. 国际呼吸杂志. 2019;(21):1604-1605-1606-1607-1608-1609-1610-1611-1612-1613-1614-1615.
- [Background] Liu M, Klein E, Hubbell E, et al. Plasma cell-free DNA (cfDNA) assays for early multi-cancer detection: the circulating cell-free genome atlas (CCGA) study. Annals of Oncology. 2018;29:viii14.
- [Background] Liu MC, Oxnard GR, Klein EA, Swanton C, Seiden MV; CCGA Consortium. Sensitive and specific multi-cancer detection and localization using methylation signatures in cell-free DNA. Ann Oncol. 2020 Jun;31(6):745-759. doi: 10.1016/j.annonc.2020.02.011. Epub 2020 Mar 30. PMID 33506766
- [Background] Eissa MAL, Lerner L, Abdelfatah E, Shankar N, Canner JK, Hasan NM, Yaghoobi V, Huang B, Kerner Z, Takaesu F, Wolfgang C, Kwak R, Ruiz M, Tam M, Pisanic TR 2nd, Iacobuzio-Donahue CA, Hruban RH, He J, Wang TH, Wood LD, Sharma A, Ahuja N. Promoter methylation of ADAMTS1 and BNC1 as potential biomarkers for early detection of pancreatic cancer in blood. Clin Epigenetics. 2019 Apr 5;11(1):59. doi: 10.1186/s13148-019-0650-0. PMID 30953539
- [Background] Singh N, Rashid S, Rashid S, Dash NR, Gupta S, Saraya A. Clinical significance of promoter methylation status of tumor suppressor genes in circulating DNA of pancreatic cancer patients. J Cancer Res Clin Oncol. 2020 Apr;146(4):897-907. doi: 10.1007/s00432-020-03169-y. Epub 2020 Mar 7. PMID 32146565
- [Background] Henriksen SD, Stubbe BE, Madsen PH, Johansen JS, Jensen BV, Hansen CP, Johansen MN, Pedersen IS, Krarup H, Thorlacius-Ussing O. Cell-free DNA promoter hypermethylation as a diagnostic marker for pancreatic ductal adenocarcinoma - An external validation study. Pancreatology. 2021 Sep;21(6):1081-1091. doi: 10.1016/j.pan.2021.05.003. Epub 2021 May 8. PMID 33994313
- [Background] Shen Q, Polom K, Williams C, de Oliveira FMS, Guergova-Kuras M, Lisacek F, Karlsson NG, Roviello F, Kamali-Moghaddam M. A targeted proteomics approach reveals a serum protein signature as diagnostic biomarker for resectable gastric cancer. EBioMedicine. 2019 Jun;44:322-333. doi: 10.1016/j.ebiom.2019.05.044. Epub 2019 May 28. PMID 31151932
- [Background] Yu J, Ploner A, Kordes M, Lohr M, Nilsson M, de Maturana MEL, Estudillo L, Renz H, Carrato A, Molero X, Real FX, Malats N, Ye W. Plasma protein biomarkers for early detection of pancreatic ductal adenocarcinoma. Int J Cancer. 2021 Apr 15;148(8):2048-2058. doi: 10.1002/ijc.33464. Epub 2021 Jan 15. PMID 33411965
- [Background] Lindgaard SC, Sztupinszki Z, Maag E, Chen IM, Johansen AZ, Jensen BV, Bojesen SE, Nielsen DL, Hansen CP, Hasselby JP, Nielsen KR, Szallasi Z, Johansen JS. Circulating Protein Biomarkers for Use in Pancreatic Ductal Adenocarcinoma Identification. Clin Cancer Res. 2021 May 1;27(9):2592-2603. doi: 10.1158/1078-0432.CCR-20-4215. Epub 2021 Mar 18. PMID 33737308
- [Background] Fehlmann T, Kahraman M, Ludwig N, Backes C, Galata V, Keller V, Geffers L, Mercaldo N, Hornung D, Weis T, Kayvanpour E, Abu-Halima M, Deuschle C, Schulte C, Suenkel U, von Thaler AK, Maetzler W, Herr C, Fahndrich S, Vogelmeier C, Guimaraes P, Hecksteden A, Meyer T, Metzger F, Diener C, Deutscher S, Abdul-Khaliq H, Stehle I, Haeusler S, Meiser A, Groesdonk HV, Volk T, Lenhof HP, Katus H, Balling R, Meder B, Kruger R, Huwer H, Bals R, Meese E, Keller A. Evaluating the Use of Circulating MicroRNA Profiles for Lung Cancer Detection in Symptomatic Patients. JAMA Oncol. 2020 May 1;6(5):714-723. doi: 10.1001/jamaoncol.2020.0001. PMID 32134442
- [Background] So JBY, Kapoor R, Zhu F, Koh C, Zhou L, Zou R, Tang YC, Goo PCK, Rha SY, Chung HC, Yoong J, Yap CT, Rao J, Chia CK, Tsao S, Shabbir A, Lee J, Lam KP, Hartman M, Yong WP, Too HP, Yeoh KG. Development and validation of a serum microRNA biomarker panel for detecting gastric cancer in a high-risk population. Gut. 2021 May;70(5):829-837. doi: 10.1136/gutjnl-2020-322065. Epub 2020 Oct 7. PMID 33028667
- [Background] Haber DA, Velculescu VE. Blood-based analyses of cancer: circulating tumor cells and circulating tumor DNA. Cancer Discov. 2014 Jun;4(6):650-61. doi: 10.1158/2159-8290.CD-13-1014. Epub 2014 May 6. PMID 24801577
- [Background] Dawson SJ, Tsui DW, Murtaza M, Biggs H, Rueda OM, Chin SF, Dunning MJ, Gale D, Forshew T, Mahler-Araujo B, Rajan S, Humphray S, Becq J, Halsall D, Wallis M, Bentley D, Caldas C, Rosenfeld N. Analysis of circulating tumor DNA to monitor metastatic breast cancer. N Engl J Med. 2013 Mar 28;368(13):1199-209. doi: 10.1056/NEJMoa1213261. Epub 2013 Mar 13. PMID 23484797
- [Background] Abbosh C, Birkbak NJ, Wilson GA, Jamal-Hanjani M, Constantin T, Salari R, Le Quesne J, Moore DA, Veeriah S, Rosenthal R, Marafioti T, Kirkizlar E, Watkins TBK, McGranahan N, Ward S, Martinson L, Riley J, Fraioli F, Al Bakir M, Gronroos E, Zambrana F, Endozo R, Bi WL, Fennessy FM, Sponer N, Johnson D, Laycock J, Shafi S, Czyzewska-Khan J, Rowan A, Chambers T, Matthews N, Turajlic S, Hiley C, Lee SM, Forster MD, Ahmad T, Falzon M, Borg E, Lawrence D, Hayward M, Kolvekar S, Panagiotopoulos N, Janes SM, Thakrar R, Ahmed A, Blackhall F, Summers Y, Hafez D, Naik A, Ganguly A, Kareht S, Shah R, Joseph L, Marie Quinn A, Crosbie PA, Naidu B, Middleton G, Langman G, Trotter S, Nicolson M, Remmen H, Kerr K, Chetty M, Gomersall L, Fennell DA, Nakas A, Rathinam S, Anand G, Khan S, Russell P, Ezhil V, Ismail B, Irvin-Sellers M, Prakash V, Lester JF, Kornaszewska M, Attanoos R, Adams H, Davies H, Oukrif D, Akarca AU, Hartley JA, Lowe HL, Lock S, Iles N, Bell H, Ngai Y, Elgar G, Szallasi Z, Schwarz RF, Herrero J, Stewart A, Quezada SA, Peggs KS, Van Loo P, Dive C, Lin CJ, Rabinowitz M, Aerts HJWL, Hackshaw A, Shaw JA, Zimmermann BG; TRACERx consortium; PEACE consortium; Swanton C. Phylogenetic ctDNA analysis depicts early-stage lung cancer evolution. Nature. 2017 Apr 26;545(7655):446-451. doi: 10.1038/nature22364. PMID 28445469
- [Background] Cree IA, Uttley L, Buckley Woods H, Kikuchi H, Reiman A, Harnan S, Whiteman BL, Philips ST, Messenger M, Cox A, Teare D, Sheils O, Shaw J; UK Early Cancer Detection Consortium. The evidence base for circulating tumour DNA blood-based biomarkers for the early detection of cancer: a systematic mapping review. BMC Cancer. 2017 Oct 23;17(1):697. doi: 10.1186/s12885-017-3693-7. PMID 29061138
- [Background] Cohen JD, Javed AA, Thoburn C, Wong F, Tie J, Gibbs P, Schmidt CM, Yip-Schneider MT, Allen PJ, Schattner M, Brand RE, Singhi AD, Petersen GM, Hong SM, Kim SC, Falconi M, Doglioni C, Weiss MJ, Ahuja N, He J, Makary MA, Maitra A, Hanash SM, Dal Molin M, Wang Y, Li L, Ptak J, Dobbyn L, Schaefer J, Silliman N, Popoli M, Goggins MG, Hruban RH, Wolfgang CL, Klein AP, Tomasetti C, Papadopoulos N, Kinzler KW, Vogelstein B, Lennon AM. Combined circulating tumor DNA and protein biomarker-based liquid biopsy for the earlier detection of pancreatic cancers. Proc Natl Acad Sci U S A. 2017 Sep 19;114(38):10202-10207. doi: 10.1073/pnas.1704961114. Epub 2017 Sep 5. PMID 28874546
- [Background] Cohen JD, Li L, Wang Y, Thoburn C, Afsari B, Danilova L, Douville C, Javed AA, Wong F, Mattox A, Hruban RH, Wolfgang CL, Goggins MG, Dal Molin M, Wang TL, Roden R, Klein AP, Ptak J, Dobbyn L, Schaefer J, Silliman N, Popoli M, Vogelstein JT, Browne JD, Schoen RE, Brand RE, Tie J, Gibbs P, Wong HL, Mansfield AS, Jen J, Hanash SM, Falconi M, Allen PJ, Zhou S, Bettegowda C, Diaz LA Jr, Tomasetti C, Kinzler KW, Vogelstein B, Lennon AM, Papadopoulos N. Detection and localization of surgically resectable cancers with a multi-analyte blood test. Science. 2018 Feb 23;359(6378):926-930. doi: 10.1126/science.aar3247. Epub 2018 Jan 18. PMID 29348365